CLINICAL TRIAL: NCT04022252
Title: Investigation of the Effects of Photobiomodulation Applications on Orthodontic Tooth Movement
Brief Title: Investigation of the Photobiomodulation Applications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Merve Goymen, Head of Orthodontics, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 261
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Orthodontic Tooth Movement
Keywords: orthodontics; tooth movement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tooth Movement (Experimental): Canine distalization on premolar extracted patients
  Interventions: Device: Cheese dental laser; Device: OrthoPulse; Other: Placebo
- Biochemistry measurements (Experimental): biochemistry analysis of IL-8, OPG, RANKL
  Interventions: Device: Cheese dental laser; Device: OrthoPulse; Other: Placebo
- periodontal measurements (Experimental): gingival and plaque index, blooding on probing, pocket depth
  Interventions: Device: Cheese dental laser; Device: OrthoPulse; Other: Placebo

INTERVENTIONS:
Device: Cheese dental laser — 810 nm GaAlAs diode laser device
Device: OrthoPulse — 850 nm LED (light emitting diode)
Other: Placebo — 810 nm GaAlAs diode laser device

SUMMARY:
Increasing the speed of orthodontic treatment is an emerging clinical problem and therefore the evaluation of the effects of photobiomodulation applications and methods on orthodontic tooth movement is considered as an important factor.

When literature studies are examined, different studies have been performed on Laser and LED applications, however, the lack of a study that evaluates and compares the effectiveness of these methods in terms of clinical and biochemical parameters.

The aim of this study is to compare the effects of laser and LED applications on tooth movement speed and to investigate the effects of these applications on the gingival fluid IL-8, OPG, RANKL. Total of 24 patients with maxillary first-premolar extraction orthodontic treatment will be included in this study, and this study will consist of 3 groups, Laser, LED and placebo group. The laser will be applied on days 0,3,7,14,21,28,35, take impression of teeth and gingival fluid samples will be collected in these days.

LED group will be given 10 minutes LED for 30 days, taken impression and DOS samples will be collected on specified days. In the placebo group, the non-active pulse laser light will be kept in the teeth and the patients will not know which group in they are. Thus, the psychological dimension of the applications will be eliminated. Sampling will be done for the placebo group on the days determined.

The investigator's project proposal consists of a total of 5 work packages; Determination of patient groups in the 1st stage and obtaining consent forms, 2nd stage Photobiomodulation applications (laser, LED, placebo application), 3rd stage orthodontic measurement and evaluation of these measurements 3D environment, taking gingival fluid samples in the 4th stage and evaluating them biochemically. In the 5th stage, statistical analysis and evaluation of the results will be done.

The data will be evaluated with SPSS 21.0.In this study, it is tried to reduce the time spent in the orthodontic treatment to close the extraction area. In this way, it will contribute to economy and time saving in terms of all orthodontic treatment physicians and physicians. It will illuminate the application of LED device which is more advantageous in terms of cost and space gain in clinical practice of physicians.

ELIGIBILITY:
Inclusion Criteria:

* adequate oral hygiene
* Class 2 malocclusion requiring upper-premolar extraction orthodontic treatment
* lack of congenital missing teeth in upper jaw
* no systemic disease

Exclusion Criteria:

* patients who wish to discontinue treatment
* patients who cannot provide oral hygiene

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Orthodontic tooth movement Change | 1st, 3rd, 7th, 14th, 21th, 28th, 35th day
  Measurement of orthodontic tooth movement (mm)

SECONDARY OUTCOMES:
Gingival Index Change | 1st, 3rd, 7th, 14th, 21th, 28th, 35th day
  Measurements of gingival index (according to Silness&Löe) all of teeth from 6 surface. Scale ranged from 0 to 3. All data will calculated for total mouth score.
Plaque Index Change | 1st, 3rd, 7th, 14th, 21th, 28th, 35th day
  Measurements of gingival index (according to Löe&Silness) all of teeth from 6 surface. Scale ranged from 0 to 3. All data will calculated for total mouth score.
RANKL Change | 1st, 3rd, 7th, 14th, 21th, 28th, 35th day
  Analyses of RANKL level in gingival crevicular fluid. The analysis will perform via ELISA. Data will present "pg/30sn"
OPG Change | 1st, 3rd, 7th, 14th, 21th, 28th, 35th day
  Analyses of OPG in gingival crevicular fluid
IL-8 Change | 1st, 3rd, 7th, 14th, 21th, 28th, 35th day
  Analyses of IL-8 in gingival crevicular fluid
Bleeding on Probing Change | 1st, 3rd, 7th, 14th, 21th, 28th, 35th day
  Estimation of bleeding on probing. The reason for the Bleeding of Probing measurement is for the control of oral hygiene motivations in patients' follow-up.
Periodontal Pocket Depth Change | 1st, 3rd, 7th, 14th, 21th, 28th, 35th day
  Measurement of Periodontal Pocket Depth (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Gundogar, PhD, Study Chair — Gaziantep University Periodontology Department; Seyithan Taysi, Prof, Study Chair — Gaziantep University Biochemistry Department

IPD SHARING:
Plan to Share IPD: No